CLINICAL TRIAL: NCT01877473
Title: Comparison of Reverse Remodeling and PVI Versus CFAE and/or Linear Lesions and PVI for Persistent AF
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No enrollment
Sponsor: Valley Health System (Other)
Responsible Party: Principal Investigator, Jonathan Steinberg,MD, Director, Arrhythmia Institute, Valley Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VHS 12.0031
Record Dates: First submitted 2013-05-26; First posted 2013-06-13 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Persistent Atrial Fibrillation
Keywords: atrial fibrillation; persistent AF; catheter ablation; duration of 7 days to one year; with symptoms and failure of at least one antiarrhythmic drug
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reverse remodeling (Active Comparator): Pretreatment with dofetilide or sotalol and restoration of sinus rhythm followed by PVI only ablation
  Interventions: Procedure: Ablation
- Standard ablation (Active Comparator): PVI ablation with additional CFAE and/or linear LA ablation
  Interventions: Procedure: Ablation

INTERVENTIONS:
Procedure: Ablation

SUMMARY:
The hypothesis of this study is that by facilitating reverse atrial remodeling with maintenance of sinus rhythm in the weeks preceding ablation makes it feasible to perform a simple pulmonary vein isolation (PVI) with results equivalent or superior to more complex atrial ablation for patients with persistent AF.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac disorder currently affecting 2.3 million U.S. adults with an expected increase in incidence to 5.6 million by the year 2050. Randomized clinical trials have shown that ablation was superior to antiarrhythmic drug (AAD) in maintaining sinus rhythm among patients with symptomatic predominantly paroxysmal AF. However the results for catheter ablation of persistent AF is much lower and more variable, ranging between 20-80%. Moreover there is no agreed-upon standard ablation approach. Prior studies suggest that pulmonary vein isolation (PVI) alone has an unacceptably low success rate so most laboratories supplement this approach with additional lesion sets. These include complex atrial fractionated electrograms ("CAFÉ"), autonomic denervation, and linear left atrial ablation at the roof and mitral isthmus, in an empirical manner or stepwise approach. However, these strategies are time consuming and prone to proarrhythmia, namely post-ablation atrial tachycardias which can occur with an incidence ranging from < 5 to 50%.

The lower efficacy of PVI alone in persistent AF has been attributed to adverse electrical, molecular, and structural remodeling of the atria. Collectively, atrial remodeling decreases conduction velocity and the effective refractory period, and results in a shortened atrial wavelength, which increases the number and stability of reentrant wavelets. This can cause persistence of AF independent of a focal discharge. Standard PVI addresses the "focal discharge" or trigger from the PVs that initiates AF but not necessarily the underlying atrial substrate.

Based on these concepts, we hypothesized that successful atrial reverse remodeling by temporary AAD therapy would facilitate the performance of PVI alone in patients with persistent AF. The utilization of reverse remodeling to enhance the efficiency, efficacy and safety of ablation of AF has not been tested in a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic persistent AF
* Failure of class I antiarrhythmic drug or amiodarone to control AF

Exclusion Criteria:

* Previous proarrhythmia to class III AAD including excessive QT prolongation or torsade-de-pointes
* Previous AF ablation procedure
* Congestive heart failure (NYHA III-IV functional class)
* Left ventricle ejection fraction less than 35%
* Left atrial diameter >55 mm
* Unwillingness to participate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Freedom of atrial fibrillation/flutter | One year

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Steinberg, MD, Principal Investigator — Valley Health System/Columbia University
Locations (1):
- Valley Hospital, Ridgewood, New Jersey, United States